CLINICAL TRIAL: NCT01395771
Title: Effects of a Phone Call Intervention to Promote HAART Adherence in Baoshan, China
Brief Title: Effects of a Phone Call Intervention to Promote HAART Adherence
Acronym: EPCIPHA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baoshan Prefecture Center for Disease Control and Prevention (Other Government)
Collaborators: Prince of Songkla University (Other)
Responsible Party: Director of Weibin Zheng, Baoshan Prefecture Center for Disease Control and Prevention
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: BSCDC2011HIV/AIDS; BSWSJ2011HIV/AIDS (Other Grant/Funding Number: Grantor)
Record Dates: First submitted 2011-06-18; First posted 2011-07-18 (Estimated); Last update posted 2011-07-18 (Estimated); Status verified 2011-07

CONDITIONS: Medication Adherence
Keywords: Effect; Phone call; Intervention; Promote; HAART adherence
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Phone call (Experimental): New cases and old cases will be randomly categorized into two groups,respectively,one is phone call intervention group, the other is no phone call intervention group.
  Interventions: Behavioral: Phone call intervention, no phone call intervention

INTERVENTIONS:
Behavioral: Phone call intervention, no phone call intervention — Biweekly phone call intervention +routine service will be assigned to intervention group of new cases and old cases. Only routine service will be assigned to the control group of abovementioned two kind of cases.

SUMMARY:
The adherence rate (95%) to HAART in the intervention group which receives a phone call will be higher than that(75%)of control group which does not receive a phone call.

DETAILED DESCRIPTION:
According to above eligibility criteria, getting two eligible group patients, one which are patients newly required HAART (new cases) and the other who have received HAART for 1-3 years(old cases). All eligible patients in each group will be randomly assigned to intervention and control group by block randomization. Among of them, one group with a phone call intervention, the other without. New cases will be followed up for 3 months and study outcomes will be assessed at the baseline and the 2nd week, the 1st month and 2nd month, and the 3rd month. For the old cases, study outcomes will be assessed only at the baseline survey and at the 3rd month.

ELIGIBILITY:
Inclusion criteria:

* Chinese patients with HIV/AIDS aged ≥ 18 years and for the newly required HAART patients, mainly based on their CD4 < 350 cells/mm3. But irrespective of CD4 cells for old patients who are under treatment for 1-3 years.

Exclusion criteria:

* Patients who have the inability to communicate at the beginning of study and who haven't got opportunistic infection(this item is only for new cases), who are non-Baoshan registered residence, who are foreigners, prisoners and pregnants, who have no mobile phone.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2011-05; Primary Completion 2011-09 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline HAART adherence within 3 months | HAART adherence for new cases will be assessed at the 2nd week, the 1st month and 2nd month, and the 3rd month follow-up. For old cases HAART adherence will be assessed only at the baseline survey and the 3rd month follow-up
  Adherence will be measured at different time points within 3 months follow-up (study period)

SECONDARY OUTCOMES:
Change from baseline quality of life within 3 months | Quality of life for new cases will be assessed at the baseline survey and the 2nd week, the 1st month and 2nd month, and the 3rd month. For old cases quality of life will be assessed only at the baseline survey and the end of the 3rd month
  Quality of life will be measured at different time points within 3 months study periods
CD4 cell counts | CD4 will be measured at the baseline survey and the 3rd month follow-up
  CD4 cell counts will be measured only at baseline survey and after 3 months
Number of patients with side effects | Number of side effects for new cases will be assessed at the 2nd week, the 1st month and 2nd month, and the 3rd month follow-up. For old cases the number of side effects will be assessed only at the baseline survey and the 3rd month follow-up
  The number of side effects will be measured at different time points within 3 months follow-up period
Number of opportunistic infection within 3 months | Number of opportunistic infection for new cases will be assessed at the 2nd week, the 1st month and 2nd month, and the 3rd month follow-up. For old cases number of that will be assessed only at the baseline and the 3rd month follow-up
  Number of opportunistic infection will be measured at different time points within 3 months follow-up period(study period)
Mortality | Mortality will be assessed the 3rd month follow-up
  Measurement of the number of change of mortality

CONTACTS AND LOCATIONS:
Overall Officials: Weibing Zheng, Bachelor, Study Director — Baoshan CDC
Locations (4):
- China (4):
  - Longling county hospital, Baoshan, Yunnan
  - Longyang district hospital, Baoshan, Yunnan
  - Tengchong county hospital, Baoshan, Yunnan
  - The first hospital of Baoshan Prefecture, Baoshan, Yunnan